CLINICAL TRIAL: NCT04162405
Title: Characteristics of Tinnitus in Patients With and Without Sensorineural Hearing Loss: A Matched Pair Analysis
Brief Title: Tinnitus in Patients With and Without Sensorineural Hearing Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital Sestre Milosrdnice
Other Study IDs: EP-TINN01
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Tinnitus, Subjective; Hearing Loss; Otorhinolaryngologic Diseases
Keywords: tinnitus; sensorineural hearing loss; otoacoustic emission; normacusis; questionnaire
MeSH Terms: conditions — Tinnitus; Hearing Loss; Otorhinolaryngologic Diseases; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with tinnitus and hearing loss: Patients with tinnitus and average speech-frequency tonal audiogram threshold >30 dB
  Interventions: Behavioral: Tinnitus Handicap Inventory Test
- Patients with tinnitus without hearing loss: Patients with tinnitus and average speech-frequency tonal audiogram threshold <30 dB
  Interventions: Behavioral: Tinnitus Handicap Inventory Test

INTERVENTIONS:
Behavioral: Tinnitus Handicap Inventory Test — A prospective cohort nonrandomized study of non-masked parallel paired groups. The data will be collected from an electronic database that is filled in during diagnostic processing. During the diagnostic processing, TSI and THI questionnaires will be filled in, a tone audiogram (TA) and DPOAE will be performed.
  Other Names: Distortion Product Otoacoustic Emission

SUMMARY:
The aim of this study is to evaluate hearing characteristics in patients with and without tinnitus using DPOAE and specific tinnitus severity index (TSI) and tinnitus handicap inventory (THI) questionnaires in both groups.

Purpose of the research:

Demonstrate that the characteristics of tinnitus depend on the presence and magnitude of hearing loss.

Research participants:

150 patients coming for further audiological treatment due to tinnitus. Data will be collected from an electronic database that is filled in during diagnostic processing. During the diagnostic processing, TSI and THI questionnaires will be filled in, a tone audiogram (TA) and DPOAE will be performed.

DETAILED DESCRIPTION:
Tinnitus affects 17% of the total population and as many as 33% of the elderly and is the primary symptom in 60% of patients referred for audiological treatment. Tinnitus is the perception of sound without external stimuli. Its pathophysiological basis is unknown and therefore its treatment is difficult and understanding of other disorders that occur in the auditory system is impeded. The auditory system has a complex structure that consists of the organs of Corti, the afferent and efferent conduction pathways, the cortical auditory center and the connections that allow their integration. The pathology that develops in any of these parts leads to a heightened perception of sound by unknown mechanisms. Patients can describe tinnitus in a variety of ways, such as sea noise, rapid flow, ringing, howling and whistling. The measurement of otoacoustic emissions by distortion products (DPOAE) is the main method that allows the evaluation of the mechanical activity of the cochlea in patients with tinnitus. In these patients, hyperacusis plays an important role and it can often be a precursor to tinnitus. The aim of this study is to evaluate hearing characteristics in patients with and without tinnitus using DPOAE and specific tinnitus severity index (TSI) and tinnitus handicap inventory (THI) questionnaires in both groups.

Research goal:

Identify differences in tinnitus characteristics in patients with and without significant hearing impairment.

Purpose of the research:

Demonstrate that the characteristics of tinnitus depend on the presence and magnitude of the visual hearing impairment.

Research participants:

150 patients coming for further audiological treatment due to tinnitus. The data will be collected from an electronic database that is filled in during diagnostic processing. During the diagnostic processing, TSI and THI questionnaires will be filled in, a tone audiogram (TA) and DPOAE will be made.

Research plan:

A prospective cohort nonrandomized study of non-masked parallel paired groups. When receiving patients at the Hearing and Balance Center, the inclusion criteria for admission to the study are adulthood (> 18 years), tinnitus as the primary reason for referring to diagnostic treatment, and consent to complete two on-site tinnitus questionnaires. Exclusion criteria are conductive hearing impairment and incomplete questionnaires. It is planned to evaluate the differences in tinnitus character between groups of patients with and without significant hearing impairment with respect to the objective parameters of the audiogram and DPAOE.

Primary Outcome:

Identification of key differences in subjective and objective characteristics of tinnitus in patients with and without noticeable hearing impairment.

There is no risk involved in this research.

ELIGIBILITY:
Inclusion Criteria:

* adulthood (> 18 years), tinnitus as the primary reason for referring to diagnostic processing, and consent to complete two on-site tinnitus questionnaires

Exclusion Criteria:

* conductive hearing loss and incomplete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without hearing loss suffering from tinnitus, scheduled for diagnostic in a tertiary audiological center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Establishing correlations between DPOAE, TA, and THI values | 2 hours
  Evaluating whethere there are certain characteristics of tinnitus correlated with patients with and without hearing loss

CONTACTS AND LOCATIONS:
Overall Officials: Robert Trotić, MD, PhD, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No